CLINICAL TRIAL: NCT02341547
Title: A Prospective, Observational, Non-inferiority Study to Assess the Effectiveness of a Biosimilar Epoetin Alfa in Maintaining Haemoglobin Levels in Stable 'End Stage Renal Failure' Patients on Haemodialysis
Brief Title: Effectiveness of a Biosimilar Epoetin Alfa in Stable 'End Stage Renal Failure'
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Ong Loke Meng, Consultant Nephrologist and Head of Medical Department, Penang Hospital, Malaysia
Other Study IDs: CT14-HPP-003
Record Dates: First submitted 2015-01-13; First posted 2015-01-19 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: End Stage Renal Failure; Anaemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: a Biosimilar Epoetin Alfa — End Stage Renal Failure patients stable on Eprex switched to Binocrit
  Other Names: Binocrit

SUMMARY:
This is a prospective, observational, non-inferior study in ESRF patients stable on Eprex who are switched to a Biosimilar Epoetin Alfa. Study plans to recrut 44 patients. Following recruitment, a baseline data collection of full routine laboratory test before switch to Binocrit.Primary endpoint is Mean change in haemoglobin levels at 12 weeks and Secondary endpoint is Mean change in haemoglobin levels at 6 weeks Safety endpoint will be Adverse drug reactions and serious adverse effects Analysis: Changes from baseline at Week 6 and Week 12 will be evaluated using paired t-test or Wilcoxon signed ranks test as appropriate. Changes in continuous variables over time were evaluated using repeated-measures analysis of variance. Patients with iron-deficiency (ferritin <100 ng/ml or transferrin saturation <20%) will be analysed separately

DETAILED DESCRIPTION:
Anaemia in CKD is associated with reduced quality of life and increased cardiovascular disease, hospitalizations, cognitive impairment, and mortality. Correcting anaemia is considered an important part of slowing or even stopping the progression of CKD. Recombinant human erythropoietins (EPO) such as epoetin alfa are erythropoiesis-stimulating agents (ESAs) that are important treatment options. The ESA that is currently used in the hospital is Eprex®, a recombinant human EPO epoetin alfa which will soon be replaced by Binocrit®, a biosimilar ESA approved by the European Medicines Agency (EMA). We want to see whether maintenance of haemoglobin in stable ESRF patients would be affected by this switch in real life practice in the Malaysian population.

This is a prospective, observational, non-inferiority study in ESRF patients stable on Eprex who are switched to a Bio similar Epoetin Alfa .

Study population will be 44 End stage renal failure patients from Penang and Seberang Jaya hospital.Following recruitment, a baseline data collection of full routine laboratory test before switch to a Bio similar Epoetin Alfa .Primary endpoint is Mean change in haemoglobin levels at 6 weeks and Secondary endpoint is Mean change in haemoglobin levels at 12 weeks Safety endpoint will be Adverse drug reactions and serious adverse effects Analysis: Changes from baseline at Week 6 and Week 12 will be evaluated using paired t-test or Wilcoxon signed ranks test as appropriate. Changes in continuous variables over time were evaluated using repeated-measures analysis of variance. Patients with iron-deficiency (ferritin <100 ng/ml or transferrin saturation <20%) will be analysed separately

ELIGIBILITY:
Inclusion Criteria:

1. End Stage Renal Failure (ESRF) patients on 3x per week HD for at least 6 months who are planned for conversion to Binocrit
2. Stable dose of Eprex and iron for at least 3 months
3. No active bleeding

Exclusion Criteria:

1. Allergy to erythropoietin
2. Bone marrow disorder
3. Acute/chronic bleeding
4. Acute illness requiring hospitalization within the last 3 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: End Stage Renal Failure (ESRF) patients stable on Eprex who are switched over to Binocrit
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in haemoglobin levels | 12 weeks

SECONDARY OUTCOMES:
Adverse drug reactions and serious adverse effects | 12 weeks
  It is a composite end point

CONTACTS AND LOCATIONS:
Overall Officials: Ong Loke Meng, FRCS, Principal Investigator — Penang Hospital